CLINICAL TRIAL: NCT03276559
Title: Enhancing & Mobilizing the POtential for Wellness & Emotional Resilience Among Surrogate Decision-Makers of ICU Patients
Acronym: EMPOWER
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Weill Medical College of Cornell University (Other)
Collaborators: New York Hospital Queens (Other); Memorial Sloan Kettering Cancer Center (Other); National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1610017622; R21CA218313 (NIH)
Record Dates: First submitted 2017-08-15; First posted 2017-09-08 (Actual); Results first posted 2024-08-20 (Actual); Last update posted 2024-08-20 (Actual); Status verified 2024-07

CONDITIONS: Critical Illness; Communication Disabilities
Keywords: critically ill; ICU; uncommunicative; caregivers; surrogate; decision-making
MeSH Terms: conditions — Critical Illness; Communication Disorders

STUDY DESIGN:
Intervention Model Description: Open trial pilot and manual refinement phase followed by randomized controlled trial. Due to the COVID-19 pandemic, we included the open-trial COVID-19 phase to adjust to new circumstances. We resumed the randomized controlled trial once it was safe to do so.
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Randomized controlled trial EMPOWER arm (Experimental): The EMPOWER arm includes six 15 minute modules delivered in a 1-on-1 format with the same interventionist, and 2 boosters (approximately 45 minutes each) conducted by phone.
  Subjects who meet eligibility criteria will receive up to 4 sequential assessments before and after the EMPOWER intervention within 3 months conducted in person and by phone.
  Interventions: Behavioral: EMPOWER
- Randomized controlled trial Enhanced usual care arm (Placebo Comparator): The usual care arm indicates regular ICU support for informal caregivers (i.e. social work, chaplaincy) as recorded in the patient's medical record, a general information packet for informal caregivers, and a site-specific resource list.
  Subjects who meet eligibility criteria will receive up to 4 sequential assessments before and after the usual care within 3 months conducted in person and by phone.
  Interventions: Other: Enhanced Usual Care
- Open trial COVID-19 phase arm (Experimental): The COVID-19 open trial phase arm did not include randomization or control arm. All participants received the EMPOWER intervention. Assessments will occur pre-intervention, immediately post-intervention, and then 1-month and 3-months from post-intervention assessment.
  Interventions: Behavioral: EMPOWER

INTERVENTIONS:
Behavioral: EMPOWER — EMPOWER is a manualized treatment delivered based in cognitive behavioral and acceptance and commitment therapies delivered by a trained mental health professional that utilizes breathing and grounding exercises, mindfulness meditation, psychoeducation, imaginal dialogue with the patient, and coping rehearsal techniques.
  The total amount of time EMPOWER intervention is about 90 minutes, about 15 minutes each module. It can either be administered in one session or many sessions to accommodate the dynamic nature of ICU, and has two booster follow-up calls (roughly 45 minutes each) in the month following initial treatment.
  Arms: Open trial COVID-19 phase arm; Randomized controlled trial EMPOWER arm
Other: Enhanced Usual Care — Enhanced usual care consists of standard ICU psychosocial support for caregivers like social work, chaplaincy, or palliative care team visits as charted in the patient's medical record. Participants assigned to EUC will also receive a general information guide for caregivers as well as a site-specific list of caregiver resources.
  Arms: Randomized controlled trial Enhanced usual care arm

SUMMARY:
Intensive Care Units (ICU) are stressful places where life-and-death medical decisions are made and patients' surrogate decision-makers are exposed to potentially traumatic experiences. As the number of life-prolonging procedures administered to the patient rises, the patient's quality of life falls. Thus, interventions to improve the quality of life and care of ICU patients are needed.

EMPOWER is a cognitive-behavioral, acceptance-based intervention for patient surrogate decision-makers to reduce experiential avoidance of unpleasant thoughts and feelings related to thinking about patient death. By reducing surrogate's experiential avoidance, EMPOWER removes a barrier to advance care planning. EMPOWER aims to improve patient quality of life through enhancing value-directed end-of-life care while also empowering surrogates to cope with a loved one's potential impending death and adjust following the patient's ICU death or discharge. Specifically, investigators aim to:

* 1: Develop EMPOWER for surrogate decision-makers of critically ill patients who are at risk of becoming incapacitated or are currently unable to communicate in the ICU. Key informants, including bereaved ICU patient caregivers and clinicians, will be asked to evaluate the EMPOWER intervention manual to increase its potential tolerability, acceptability and efficacy.
* 2: Determine feasibility, tolerability, acceptability, and preliminary effects of EMPOWER on surrogate mental health.
* 3: Estimate the effects of EMPOWER on patient outcomes in the months following the ICU admission.

Hypothesis 1: Surrogate decision-makers who receive EMPOWER will have significantly lower levels of peritraumatic distress when compared to usual care condition at post intervention assessment (T2).

Hypothesis 2: Patients whose surrogates receive EMPOWER will have more value-concordant care, better quality of life, and better quality of death.

EMPOWER was first evaluated though a single site open trial (n=10). All 10 participants in the open trial phase received EMPOWER. Feedback from clinicians, bereaved stakeholders and results from the open trial were then used to refine the intervention and launch a multi-center randomized controlled trial to examine clinical superiority of EMPOWER to enhanced usual care. In order to adapt to restrictions in ICU visitation and meet the needs of family caregivers impacted by the COVID-19 pandemic, we then launched a second single arm open trial and paused recruitment for the RCT. All participants recruited during the open trial COVID-19 phase received EMPOWER. Beginning in August 2021, we resumed the RCT portion of the trial to meet the initial recruitment goals of the study (total n of RCT & COVID-19 open trial=60).

DETAILED DESCRIPTION:
Aggressive care in Intensive Care Units (ICUs) has been shown to impair the quality of life of patients with advanced cancer and to increase the risk of Posttraumatic Stress Disorder (PTSD) among the family and friends who serve as informal caregivers. Although ICU stays are established indicators of low quality end-of-life (EoL) cancer care, a large, growing number of cancer patients - over 1 in 4 -- are being admitted to the ICU in the last month of life. Even within the ICU, investigators find that as the number of life-prolonging procedures administered to the patient rises, the patient's quality of life falls. Thus, interventions to reduce the suffering and to improve the quality of life and care of ICU cancer patients are needed.

As described above, suffering is not confined to the patient. Informal caregivers of cancer patients in the ICU also suffer. In our "Severity of Suffering" (SoS) study, which examined dying cancer patients' quality of life in the ICU, nurses indicated that 53% of the patients' caregivers were acutely distressed. The nurses also reported that 43% of the patient's caregivers had unrealistic expectations for the patient's recovery and that 41% insisted that the patient receive futile, burdensome care (e.g., resuscitation). Over 85% of these patients were unable to communicate, which resulted in the need for grieving, potentially traumatized caregivers to serve as the patient's surrogate decision-maker and make life-and-death decisions for a critically ill, uncommunicative patient. Additionally, caregivers of patients who die in the ICU are also at elevated risk of posttraumatic stress disorder (PTSD) in the months that follow the potentially traumatic ICU "exposures". These findings indicate a compelling need to address the varying mental health needs of informal caregivers and surrogate decision-makers of patients in the ICU from admission to after discharge, as well as to provide them with resources to clarify and inform the decision-making process regarding care for patients who are unable to communicate.

To address these needs, we have developed and will refine and evaluate EMPOWER, a mental health intervention for surrogate decision-makers of ICU patients who are at risk of becoming incapacitated or are currently unable to make medical decisions. Delivered by a trained mental health professional in the ICU setting, EMPOWER is a cognitive-behavioral, acceptance-based intervention designed to reduce "experiential avoidance" of unpleasant thoughts and feelings related to thinking about the patient's death and to provide active strategies for coping with peritraumatic distress and anticipatory grief. Additionally, by reducing surrogates' experiential avoidance, EMPOWER removes a barrier to advanced care planning and promotes the receipt of EoL care consistent with patient values. In this way, EMPOWER aims to facilitate EoL care that enhances patient quality of life while also empowering surrogates to cope with a loved one's potential impending death and adjust following the patient's ICU death or discharge.

This study is designed to obtain information on its feasibility, tolerability, acceptability, and preliminary effect size estimates to inform the planning of a larger, efficacy randomized controlled trial (RCT). In order to develop the RCT, the first 10 surrogate decision-makers were enrolled in an open trial to receive EMPOWER. In addition, during the manual refinement phase, up to 15 stakeholders (bereaved caregivers of ICU patients) were interviewed after reviewing the EMPOWER intervention manual. We then began a pilot RCT, randomizing surrogate decision-makers to receive either EMPOWER or enhanced usual care using a block-randomization strategy to determine condition assignment. In light of restrictions on recruitment and increased needs of surrogates during the COVID-19 pandemic, we paused the RCT portion of this trial and we recruited for a second open trial only administering EMPOWER. 60 surrogate-patient dyads were enrolled between the RCT and COVID-19 open trial. In August 2021, we resumed the RCT trial of the study. We resumed in person recruitment and randomization of participants to EMPOWER or EUC. Including the first open trial, we will enroll a total of 70 surrogate decision-makers of 70 current patients from the intensive care units at New York Presbyterian-Weill Cornell, New York Presbyterian-Queens, and Memorial Sloan Kettering Cancer Center. Research staff will regularly contact ICU physicians in person or by email and/or screen patient charts to identify eligible candidates based on the inclusion criteria.

Surrogates will be consented and screened. Those who score above 5 on either item measuring anxiety in the McGill Quality of Life Scale, or with a summed score of at least 8 on the first two items of the Partner Dependency Scale (PDS) will be randomized to receive EMPOWER or usual care in the RCT, or solely assigned to receive the intervention in the pilot trials. Surrogates will be assessed pre-intervention/baseline (Time point 1, T1), post-intervention (within a week of the surrogate's completion of the baseline assessment) (Time point 2, T2), 1-month post-T2 (Time point 3, T3), and 3-months post-T2(Time point 4, T4). Surrogates will be assigned to either control (usual care) or intervention group using block randomization in the RCT, and solely to EMPOWER in open trials.

EMPOWER is based on well-established cognitive-behavioral techniques that aim to promote the expression and understanding of a person's emotional reactions. The EMPOWER interventionist will be compassionate and attempt to teach subjects tools for remaining present-focused, validate participants' experience, explore participants' loved ones' and participants' own wishes, values and decision challenges, increase subjects acceptance and sense of permission to experience challenging emotions, and prepare participants for future distressing situations. Enhanced usual care will consist of a surrogate's interactions with social support services in the ICU as documented in the patient's medical chart, referrals for current site-specific resources for informal caregivers, and a packet providing general information and tips on serving as an informal caregiver.

HLM modeling will determine differences between surrogates and patients assigned to EMPOWER vs. enhanced usual care. The primary outcome is post-intervention (T2) differences on a measure of peritraumatic distress. Secondary outcomes are differences on measures of prolonged grief disorder, PTSD and experiential avoidance at one-month (T3) and three-month (T4) follow up from T2. Exploratory outcomes for surrogates are differences in reported symptoms of anxiety, depression, and decision regret at one-month (T3) and three-month (T4) follow up from T2. Exploratory outcomes for patients are differences in surrogate-reported quality of life, quality of death, and value concordant care. HLM models will include covariates, either as fixed-effect or time-varying, if those variables are found to be significantly statistically associated with both intervention assignment and the outcome examined.

Following a review of the open trial pilot data and stakeholder feedback to evaluate our intervention targets, assessments and the primary outcome in the RCT were revised to target the effects of the EMPOWER intervention on peri (rather than post) traumatic stress.

ELIGIBILITY:
Inclusion criteria for stakeholders:

1. Bereaved family caregivers of patients treated in the ICU identified by referring clinicians and through support groups, clinics, and word of mouth
2. Clinicians with expertise in mental health care and/or critical care including but not limited to nurses, nurse practitioners, social workers, psychologists, psychiatrists, hospital chaplains, and physicians

Inclusion criteria for open trial participants:

1. Patients (>21 years) who cannot communicate and decide on treatments, who during the course of their current hospital stay were admitted to an ICU/step-down unit, and whose ICU physicians or fellows would not be surprised if the patient did not survive more than 3 months
2. Surrogate decision-makers whom ICU physicians or fellows indicate as the designated health care proxy or decision-making patient surrogates, or who are listed as such in the patient's medical charts
3. Surrogate decision-makers must speak English
4. Surrogate decision-makers must either meet the threshold for a high degree of emotional dependence (PDS 18 score >8) on the patient or on the McGill Quality of Life Scale19 items (either anxiety item score>5).

Inclusion criteria for adult pilot RCT participants:

1. Patients (>18 years) who during the course of their current hospital stay were admitted to an ICU/step-down unit
2. Surrogate decision-makers whom ICU physicians or fellows indicate as the designated health care proxy or decision-making patient surrogates, or who are listed as such in the patient's medical charts or by self-report of the surrogate
3. Surrogate decision-makers must speak English
4. Surrogate decision-makers must either meet the threshold for a high degree of emotional dependence (PDS 18 score >8) on the patient or on the McGill Quality of Life Scale 19 items (either anxiety item score>5).
5. Surrogate decision-makers who do not meet criterion #4 but are identified by clinical staff as distressed and whom clinical staff believe would benefit from the intervention.

Inclusion criteria child pilot RCT/COVID-19 Open Trial participants:

1. Patients below the age of 18 who have spent at least 3 days in a pediatric intensive care unit
2. Surrogate decision-makers whom ICU physicians or fellows indicate as the designated health care proxy or decision-making patient surrogates, or who are listed as such in the patient's medical charts or by self-report of the surrogate, or are parents of the patient
3. Surrogate decision-makers must speak English

Inclusion criteria for adult open trial COVID-19 participants:

1. Patients (>18 years) who during the course of their current hospital stay were admitted to an ICU/step-down unit
2. Surrogate decision-makers whom a member of the patient's care team indicate as the designated health care proxy or decision-making patient surrogates, or who are listed as such in the patient's medical charts
3. Surrogate decision-makers must speak English
4. Surrogate decision-makers must either meet the threshold for a high degree of emotional dependence (PDS 18 score >8) on the patient or on the McGill Quality of Life Scale items (either anxiety item score>5).
5. Surrogate decision-makers who do not meet criterion #4 but are identified by clinical staff as distressed and whom clinical staff believe would benefit from the intervention.

Exclusion criteria for all arms:

Patients and surrogate decision-makers who do not meet the eligibility criteria or surrogate decision-makers who endorse suicidal ideation in the past month based on responses to the Columbia Suicide Severity Rating Scale.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 63 (Actual)
Dates: Start 2017-07-12 (Actual); Primary Completion 2023-05-22 (Actual); Study Completion 2023-05-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Holly G Prigerson, Ph. D., Principal Investigator — Weill Medical College of Cornell University
Locations (3):
- United States (3):
  - NewYork-Presbyterian Queens, Flushing, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - NewYork-Presbyterian Weill Cornell Medicine, New York, New York

REFERENCES:
- [Background] Wright AA, Zhang B, Ray A, Mack JW, Trice E, Balboni T, Mitchell SL, Jackson VA, Block SD, Maciejewski PK, Prigerson HG. Associations between end-of-life discussions, patient mental health, medical care near death, and caregiver bereavement adjustment. JAMA. 2008 Oct 8;300(14):1665-73. doi: 10.1001/jama.300.14.1665. PMID 18840840
- [Background] Zhang B, Nilsson ME, Prigerson HG. Factors important to patients' quality of life at the end of life. Arch Intern Med. 2012 Aug 13;172(15):1133-42. doi: 10.1001/archinternmed.2012.2364. PMID 22777380
- [Background] Gamez W, Chmielewski M, Kotov R, Ruggero C, Watson D. Development of a measure of experiential avoidance: the Multidimensional Experiential Avoidance Questionnaire. Psychol Assess. 2011 Sep;23(3):692-713. doi: 10.1037/a0023242. PMID 21534697
- [Background] Prigerson HG, Shear MK, Jacobs SC, Reynolds CF 3rd, Maciejewski PK, Davidson JR, Rosenheck R, Pilkonis PA, Wortman CB, Williams JB, Widiger TA, Frank E, Kupfer DJ, Zisook S. Consensus criteria for traumatic grief. A preliminary empirical test. Br J Psychiatry. 1999 Jan;174:67-73. doi: 10.1192/bjp.174.1.67. PMID 10211154
- [Background] Mack JW, Weeks JC, Wright AA, Block SD, Prigerson HG. End-of-life discussions, goal attainment, and distress at the end of life: predictors and outcomes of receipt of care consistent with preferences. J Clin Oncol. 2010 Mar 1;28(7):1203-8. doi: 10.1200/JCO.2009.25.4672. Epub 2010 Feb 1. PMID 20124172
- [Background] Garrido MM, Prigerson HG. The end-of-life experience: modifiable predictors of caregivers' bereavement adjustment. Cancer. 2014 Mar 15;120(6):918-25. doi: 10.1002/cncr.28495. Epub 2013 Dec 2. PMID 24301644
- [Background] Wright AA, Keating NL, Balboni TA, Matulonis UA, Block SD, Prigerson HG. Place of death: correlations with quality of life of patients with cancer and predictors of bereaved caregivers' mental health. J Clin Oncol. 2010 Oct 10;28(29):4457-64. doi: 10.1200/JCO.2009.26.3863. Epub 2010 Sep 13. PMID 20837950
- [Background] Siegel MD, Hayes E, Vanderwerker LC, Loseth DB, Prigerson HG. Psychiatric illness in the next of kin of patients who die in the intensive care unit. Crit Care Med. 2008 Jun;36(6):1722-8. doi: 10.1097/CCM.0b013e318174da72. PMID 18520637
- [Background] Curtis JR, Back AL, Ford DW, Downey L, Shannon SE, Doorenbos AZ, Kross EK, Reinke LF, Feemster LC, Edlund B, Arnold RW, O'Connor K, Engelberg RA. Effect of communication skills training for residents and nurse practitioners on quality of communication with patients with serious illness: a randomized trial. JAMA. 2013 Dec 4;310(21):2271-81. doi: 10.1001/jama.2013.282081. PMID 24302090
- [Background] Lautrette A, Darmon M, Megarbane B, Joly LM, Chevret S, Adrie C, Barnoud D, Bleichner G, Bruel C, Choukroun G, Curtis JR, Fieux F, Galliot R, Garrouste-Orgeas M, Georges H, Goldgran-Toledano D, Jourdain M, Loubert G, Reignier J, Saidi F, Souweine B, Vincent F, Barnes NK, Pochard F, Schlemmer B, Azoulay E. A communication strategy and brochure for relatives of patients dying in the ICU. N Engl J Med. 2007 Feb 1;356(5):469-78. doi: 10.1056/NEJMoa063446. PMID 17267907
- [Background] Carson SS, Cox CE, Wallenstein S, Hanson LC, Danis M, Tulsky JA, Chai E, Nelson JE. Effect of Palliative Care-Led Meetings for Families of Patients With Chronic Critical Illness: A Randomized Clinical Trial. JAMA. 2016 Jul 5;316(1):51-62. doi: 10.1001/jama.2016.8474. Erratum In: JAMA. 2017 May 23;317(20):2134. doi: 10.1001/jama.2017.4298. PMID 27380343
- [Background] Azoulay E, Pochard F, Kentish-Barnes N, Chevret S, Aboab J, Adrie C, Annane D, Bleichner G, Bollaert PE, Darmon M, Fassier T, Galliot R, Garrouste-Orgeas M, Goulenok C, Goldgran-Toledano D, Hayon J, Jourdain M, Kaidomar M, Laplace C, Larche J, Liotier J, Papazian L, Poisson C, Reignier J, Saidi F, Schlemmer B; FAMIREA Study Group. Risk of post-traumatic stress symptoms in family members of intensive care unit patients. Am J Respir Crit Care Med. 2005 May 1;171(9):987-94. doi: 10.1164/rccm.200409-1295OC. Epub 2005 Jan 21. PMID 15665319
- [Background] Orsillo SM, Batten SV. Acceptance and commitment therapy in the treatment of posttraumatic stress disorder. Behav Modif. 2005 Jan;29(1):95-129. doi: 10.1177/0145445504270876. PMID 15557480
- [Background] Kentish-Barnes N, Prigerson HG. Is this bereaved relative at risk of prolonged grief? Intensive Care Med. 2016 Aug;42(8):1279-81. doi: 10.1007/s00134-015-4182-6. Epub 2015 Dec 23. No abstract available. PMID 26699916
- [Background] Higgins PC, Garrido MM, Prigerson HG. Factors Predicting Bereaved Caregiver Perception of Quality of Care in the Final Week of Life: Implications for Health Care Providers. J Palliat Med. 2015 Oct;18(10):849-57. doi: 10.1089/jpm.2015.29001.hp. Epub 2015 Jul 17. PMID 26186021
- [Background] Mouthaan J, Sijbrandij M, de Vries GJ, Reitsma JB, van de Schoot R, Goslings JC, Luitse JS, Bakker FC, Gersons BP, Olff M. Internet-based early intervention to prevent posttraumatic stress disorder in injury patients: randomized controlled trial. J Med Internet Res. 2013 Aug 13;15(8):e165. doi: 10.2196/jmir.2460. PMID 23942480
- [Background] Gartlehner G, Forneris CA, Brownley KA, Gaynes BN, Sonis J, Coker-Schwimmer E, Jonas DE, Greenblatt A, Wilkins TM, Woodell CL, Lohr KN. Interventions for the Prevention of Posttraumatic Stress Disorder (PTSD) in Adults After Exposure to Psychological Trauma [Internet]. Rockville (MD): Agency for Healthcare Research and Quality (US); 2013 Apr. Report No.: 13-EHC062-EF. Available from http://www.ncbi.nlm.nih.gov/books/NBK133344/ PMID 23658936
- [Background] Bryant RA, Mastrodomenico J, Felmingham KL, Hopwood S, Kenny L, Kandris E, Cahill C, Creamer M. Treatment of acute stress disorder: a randomized controlled trial. Arch Gen Psychiatry. 2008 Jun;65(6):659-67. doi: 10.1001/archpsyc.65.6.659. PMID 18519824
- [Background] Andrews B, Brewin CR, Stewart L, Philpott R, Hejdenberg J. Comparison of immediate-onset and delayed-onset posttraumatic stress disorder in military veterans. J Abnorm Psychol. 2009 Nov;118(4):767-77. doi: 10.1037/a0017203. PMID 19899846
- [Background] Prigerson HG, Horowitz MJ, Jacobs SC, Parkes CM, Aslan M, Goodkin K, Raphael B, Marwit SJ, Wortman C, Neimeyer RA, Bonanno GA, Block SD, Kissane D, Boelen P, Maercker A, Litz BT, Johnson JG, First MB, Maciejewski PK. Prolonged grief disorder: Psychometric validation of criteria proposed for DSM-V and ICD-11. PLoS Med. 2009 Aug;6(8):e1000121. doi: 10.1371/journal.pmed.1000121. Epub 2009 Aug 4. PMID 19652695
- [Background] Tomarken A, Holland J, Schachter S, Vanderwerker L, Zuckerman E, Nelson C, Coups E, Ramirez PM, Prigerson H. Factors of complicated grief pre-death in caregivers of cancer patients. Psychooncology. 2008 Feb;17(2):105-11. doi: 10.1002/pon.1188. PMID 17443644
- [Background] Prigerson HG, Viola M, Brewin CR, Cox C, Ouyang D, Rogers M, Pan CX, Rabin S, Xu J, Vaughan S, Gordon-Elliot JS, Berlin D, Lief L, Lichtenthal WG. Enhancing & Mobilizing the POtential for Wellness & Emotional Resilience (EMPOWER) among Surrogate Decision-Makers of ICU Patients: study protocol for a randomized controlled trial. Trials. 2019 Jul 9;20(1):408. doi: 10.1186/s13063-019-3515-0. PMID 31288829

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 81 caregivers consented. 16 were not eligible (eligibility's determined by a brief screening assessment conducted after participants sign consent form). 2 were loss to follow-up prior to sending the T1 assessment. 63 participants completed the first assessment (T1). After T1 is completed, participants are randomized to study groups. 60 caregivers were randomized because 1 patient died (patients were not considered enrolled in the study), 1 patient was discharged, and 1 was loss to follow-up.
Groups:
- Randomized Controlled Trial EMPOWER Arm: The EMPOWER arm includes six 15 minute modules delivered in a 1-on-1 format with the same interventionist, and 2 boosters (approximately 45 minutes each) conducted by phone.
  Subjects who meet eligibility criteria will receive up to 4 sequential assessments before and after the EMPOWER intervention within 3 months conducted in person and by phone.
  EMPOWER: EMPOWER is a manualized cognitive-behavioral, acceptance-based intervention delivered by a trained mental health professional that utilizes breathing and grounding exercises, mindfulness meditation, psycho-education, and imaginal dialogue with the patient and coping rehearsal techniques.
  The total amount of time EMPOWER intervention is about 90 minutes, about 15 minutes each module. It can either be administered in one session or many sessions to accommodate the dynamic nature of ICU, and has two booster follow-up calls (roughly 45 minutes each) in the month following initial treatment.
- Randomized Controlled Trial Enhanced Usual Care Arm: The usual care arm indicates regular ICU support for informal caregivers (i.e. social work, chaplaincy) as recorded in the patient's medical record, a general information packet for informal caregivers, and a site-specific resource list.
  Subjects who meet eligibility criteria will receive up to 4 sequential assessments before and after the usual care within 3 months conducted in person and by phone.
  Enhanced Usual Care: Enhanced usual care consists of standard ICU psychosocial support for caregivers like social work, chaplaincy, or palliative care team visits as charted in the patient's medical record. Participants assigned to EUC will also receive a general information guide for caregivers as well as a site-specific list of caregiver resources.
- Open Trial COVID-19 Phase Arm: The COVID-19 open trial phase arm did not include randomization or control arm. All participants received the EMPOWER intervention. Assessments will occur pre-intervention, immediately post-intervention, and then 1-month and 3-months from post-intervention assessment.
  EMPOWER: EMPOWER is a manualized cognitive-behavioral, acceptance-based intervention delivered by a trained mental health professional that utilizes breathing and grounding exercises, mindfulness meditation, psycho-education, and imaginal dialogue with the patient and coping rehearsal techniques.
  The total amount of time EMPOWER intervention is about 90 minutes, about 15 minutes each module. It can either be administered in one session or many sessions to accommodate the dynamic nature of ICU, and has two booster follow-up calls (roughly 45 minutes each) in the month following initial treatment.
- T1 Assessment: All participants that completed the first assessment (T1).
Period: T1 Assessment
Arm/Group | Randomized Controlled Trial EMPOWER Arm | Randomized Controlled Trial Enhanced Usual Care Arm | Open Trial COVID-19 Phase Arm | T1 Assessment
Started | 0 | 0 | 0 | 63
Completed | 0 | 0 | 0 | 63
Not Completed | 0 | 0 | 0 | 0
Period: Randomization
Arm/Group | Randomized Controlled Trial EMPOWER Arm | Randomized Controlled Trial Enhanced Usual Care Arm | Open Trial COVID-19 Phase Arm | T1 Assessment
Started (Please note that the 25 EMPOWER-Only subjects in the Open trial COVID-19 phase arm are different from the 17 subjects enrolled in the earlier period, and are different than the 20 subjects enrolled in the later period.) | 10 | 7 | 0 | 0
Completed | 5 | 5 | 0 | 0
Not Completed | 5 | 2 | 0 | 0
Period: EMPOWER Only
Arm/Group | Randomized Controlled Trial EMPOWER Arm | Randomized Controlled Trial Enhanced Usual Care Arm | Open Trial COVID-19 Phase Arm | T1 Assessment
Started | 0 | 0 | 23 | 0
Completed | 0 | 0 | 14 | 0
Not Completed | 0 | 0 | 9 | 0
Period: Randomization
Arm/Group | Randomized Controlled Trial EMPOWER Arm | Randomized Controlled Trial Enhanced Usual Care Arm | Open Trial COVID-19 Phase Arm | T1 Assessment
Started | 10 | 10 | 0 | 0
Completed | 5 | 6 | 0 | 0
Not Completed | 5 | 4 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Randomized Controlled Trial EMPOWER Arm: The EMPOWER arm includes six 15 minute modules delivered in a 1-on-1 format with the same interventionist, and 2 boosters (approximately 45 minutes each) conducted by phone.
  Subjects who meet eligibility criteria will receive up to 4 sequential assessments before and after the EMPOWER intervention within 3 months conducted in person and by phone.
  EMPOWER: EMPOWER is a manualized treatment delivered based in cognitive behavioral and acceptance and commitment therapies delivered by a trained mental health professional that utilizes breathing and grounding exercises, mindfulness meditation, psychoeducation, imaginal dialogue with the patient, and coping rehearsal techniques.
  The total amount of time EMPOWER intervention is about 90 minutes, about 15 minutes each module. It can either be administered in one session or many sessions to accommodate the dynamic nature of ICU, and has two booster follow-up calls (roughly 45 minutes each) in the month following initial treatment.
- Open Trial COVID-19 Phase Arm: The COVID-19 open trial phase arm did not include randomization or control arm. All participants received the EMPOWER intervention. Assessments will occur pre-intervention, immediately post-intervention, and then 1-month and 3-months from post-intervention assessment.
  EMPOWER: EMPOWER is a manualized treatment delivered based in cognitive behavioral and acceptance and commitment therapies delivered by a trained mental health professional that utilizes breathing and grounding exercises, mindfulness meditation, psychoeducation, imaginal dialogue with the patient, and coping rehearsal techniques.
  The total amount of time EMPOWER intervention is about 90 minutes, about 15 minutes each module. It can either be administered in one session or many sessions to accommodate the dynamic nature of ICU, and has two booster follow-up calls (roughly 45 minutes each) in the month following initial treatment.
- Total: Total of all reporting groups
Arm/Group | Randomized Controlled Trial EMPOWER Arm | Randomized Controlled Trial Enhanced Usual Care Arm | Open Trial COVID-19 Phase Arm | Total
Number analyzed (Participants) | 20 | 17 | 23 | 60
Age, Categorical [Count of Participants; unit: Participants] — Population: 2 participants in the Randomized Controlled Trial EMPOWER Arm have missing age data, which is why the number analyzed is 18 participants instead of 20 participants.
  Participants
    number analyzed (Participants) | 18 | 17 | 23 | 58
    <=18 years | 0 | 0 | 0 | 0
    Between 18 and 65 years | 17 | 13 | 23 | 53
    >=65 years | 1 | 4 | 0 | 5
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: 2 participants in the Randomized Controlled Trial EMPOWER Arm have missing age data, which is why the number analyzed is 18 participants instead of 20 participants.
  years
    number analyzed (Participants) | 18 | 17 | 23 | 58
    (all) | 43.635 (11.313) | 51.413 (15.705) | 42.091 (9.282) | 45.303 (12.523)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15 | 13 | 17 | 45
  Male | 5 | 4 | 6 | 15
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 5 | 4 | 7 | 16
  Not Hispanic or Latino | 14 | 10 | 15 | 39
  Unknown or Not Reported | 1 | 3 | 1 | 5
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 2 | 2 | 1 | 5
  Native Hawaiian or Other Pacific Islander | 1 | 2 | 0 | 3
  Black or African American | 3 | 2 | 6 | 11
  White | 12 | 9 | 7 | 28
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 2 | 2 | 9 | 13
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 20 | 17 | 23 | 60

OUTCOME MEASURES:

1. Primary Outcome: Change in Peritraumatic Distress Inventory
Description: Symptoms of peritraumatic distress, as measured by the Peritraumatic Distress Inventory (adapted to fit the ICU experience), will be compared between groups at post-intervention assessment (T2). The PDI consists of 13 likert-style items and total score can range from 0 to 52. Higher total scores represent greater symptom burden. Lower scores represent better outcomes.
Time Frame: At baseline (T1) and in the week following the intervention (T2)
Population: As pre-specified in the analysis plan, "Randomized Controlled Trial EMPOWER Arm" and "Open Trial COVID-19 Phase Arm" are combined because there were no procedural differences for subjects in both groups, besides the "Randomized Controlled Trial EMPOWER Arm" subjects were randomized to that group instead of the usual care group. Subjects in both the "Randomized Controlled Trial EMPOWER Arm" and "Open Trial COVID-19 Phase Arm" received the EMPOWER intervention and were thus analyzed together.
Measure: Mean (95% Confidence Interval); unit: score on a scale
Groups:
- Randomized Controlled Trial EMPOWER + Open Trial COVID-19 Phase Arm Combined: EMPOWER is a manualized cognitive-behavioral, acceptance-based intervention delivered by a trained mental health professional that utilizes breathing and grounding exercises, mindfulness meditation, psycho-education, and imaginal dialogue with the patient and coping rehearsal techniques.
  The total amount of time EMPOWER intervention is about 90 minutes, about 15 minutes each module. It can either be administered in one session or many sessions to accommodate the dynamic nature of ICU, and has two booster follow-up calls (roughly 45 minutes each) in the month following initial treatment.
- Randomized Controlled Trial Enhanced Usual Care Arm: Enhanced usual care consists of standard ICU psychosocial support for caregivers like social work, chaplaincy, or palliative care team visits as charted in the patient's medical record. Participants assigned to EUC will also receive a general information guide for caregivers as well as a site-specific list of caregiver resources.
Arm/Group | Randomized Controlled Trial EMPOWER + Open Trial COVID-19 Phase Arm Combined | Randomized Controlled Trial Enhanced Usual Care Arm
Number analyzed (Participants) | 43 | 17
score on a scale
  Pre-Intervention Time 1 | 14.6 [12.4 to 16.8] | 14.2 [10.2 to 18.3]
  Post-Intervention Time 2 | 13.0 [9.9 to 16.0] | 14.4 [9.2 to 19.5]

2. Secondary Outcome: Change in Anticipatory Grief
Description: Anticipatory grief for patients who are not deceased, as measured by the Prolonged Grief-12, will be compared between groups at baseline (T1) and in the week following the intervention (T2), one month and three months from baseline (T3 and T4)..The PG-12 consists of 12 items and total score can range from 0 to 57. Higher total scores represent greater symptom burden. Lower scores represent better outcomes.
Time Frame: At baseline (T1) and in the week following the intervention (T2), one month and three months from baseline (T3 and T4).
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Randomized Controlled Trial EMPOWER + Open Trial COVID-19 Phase Arm Combined | Randomized Controlled Trial Enhanced Usual Care Arm
Number analyzed (Participants) | 43 | 17
score on a scale
  Pre-Intervention Time 1 | 29.1 [26.4 to 31.8] | 24.8 [20.5 to 29.2]
  Post-Intervention Time 2 | 25.7 [22.8 to 28.6] | 25.4 [20.9 to 29.0]
  One Month Time 3 | 24.2 [22.1 to 26.4] | 26.5 [21.9 to 31.2]
  Three Months Time 4 | 20.3 [17.8 to 22.9] | 23.0 [19.3 to 26.7]

3. Secondary Outcome: Change in Experiential Avoidance
Description: Symptoms of experiential avoidance, as measured by the Brief Experiential Avoidance Questionnaire, will be compared between groups at baseline (T1) and in the week following the intervention (T2), one month and three months from baseline (T3 and T4). The BEAQ consists of 15 items and total score can range from 15 to 90. Higher total scores represent greater symptom burden. Lower scores represent better outcomes.
Time Frame: At baseline (T1) and in the week following the intervention (T2), one month and three months from baseline (T3 and T4).
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Randomized Controlled Trial EMPOWER + Open Trial COVID-19 Phase Arm Combined | Randomized Controlled Trial Enhanced Usual Care Arm
Number analyzed (Participants) | 43 | 17
score on a scale
  Pre-Intervention (T1) | 44.7 [40.3 to 49.1] | 44.5 [40.2 to 48.9]
  Post-Intervention (T2) | 42.2 [39.2 to 46.3] | 40.7 [34.7 to 46.7]
  One Month Time (T3) | 43.3 [39.0 to 47.7] | 48.2 [43.2 to 53.3]
  Three Months Time (T4) | 43.2 [39.0 to 47.4] | 48.2 [41.1 to 55.3]

4. Secondary Outcome: Change in Post-Traumatic Stress Disorder
Description: Symptoms of post-traumatic stress disorder, as measured by the Impact of Events Scale-Revised, will be compared between groups at baseline (T1) and in the week following the intervention (T2), one month and three months from baseline (T3 and T4). The IES-R consists of 22 items and total score can range from 0 to 88. Higher total scores represent greater symptom burden. Lower scores represent better outcomes.
Time Frame: At baseline (T1) and in the week following the intervention (T2), one month and three months from baseline (T3 and T4).
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Randomized Controlled Trial EMPOWER + Open Trial COVID-19 Phase Arm Combined | Randomized Controlled Trial Enhanced Usual Care Arm
Number analyzed (Participants) | 43 | 17
score on a scale
  Pre-Intervention (T1) | 29.9 [25.2 to 34.5] | 24.6 [15.5 to 33.8]
  Post-Intervention (T2) | 23.1 [17.7 to 28.5] | 25.8 [16.7 to 34.9]
  One Month Time (T3) | 24.3 [18.3 to 30.2] | 29.8 [21.0 to 38.7]
  Three Months Time (T4) | 16.0 [12.1 to 19.8] | 22.1 [14.5 to 29.6]

5. Other Pre Specified Outcome: Change in Anxiety
Description: Symptoms of anxiety, as measured by the state scale of the State-Trait Anxiety Scale, will be compared between groups at baseline (T1) and in the week following the intervention (T2), one month and three months from baseline (T3 and T4).The STAI-Y state scale consists of 20 items and total score can range from 20 to 80. Higher total scores represent greater symptom burden. Lower scores represent better outcomes.
Time Frame: At baseline (T1) and in the week following the intervention (T2), one month and three months from baseline (T3 and T4).
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Randomized Controlled Trial EMPOWER + Open Trial COVID-19 Phase Arm Combined | Randomized Controlled Trial Enhanced Usual Care Arm
Number analyzed (Participants) | 43 | 17
score on a scale
  Pre-Intervention Time 1 | 40.6 [38.3 to 42.9] | 38.8 [35.4 to 42.3]
  Post-Intervention Time 2 | 37.0 [34.5 to 39.6] | 37.4 [33.4 to 41.3]
  One Month Time (T3) | 36.2 [32.9 to 38.5] | 35.4 [32.1 to 38.7]
  Three Month Time (T4) | 35.2 [32.3 to 38.1] | 32.2 [28.1 to 36.4]

6. Other Pre Specified Outcome: Change in Depression
Description: Symptoms of depression, as measured by the Patient Health Questionnaire - 9 , will be compared between groups at baseline (T1), one month and three months from baseline (T3 and T4).. The PHQ-9 consists of 9 items and total score can range from 0 to 27. Higher total scores represent greater symptom burden. Lower scores represent better outcomes.
Time Frame: At baseline (T1), one month and three months from baseline (T3 and T4).
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Randomized Controlled Trial EMPOWER + Open Trial COVID-19 Phase Arm Combined | Randomized Controlled Trial Enhanced Usual Care Arm
Number analyzed (Participants) | 43 | 17
score on a scale
  Pre-Intervention Time 1 | 8.9 [6.7 to 10.4] | 6.8 [4.3 to 9.2]
  One Month Time 3 | 6.9 [5.9 to 12.5] | 9.2 [5.9 to 12.5]
  Three Months Time 4 | 7.6 [5.6 to 9.6] | 8.2 [5.4 to 11.1]

7. Other Pre Specified Outcome: Change in Decision Regret
Description: Decision regret, as measured by the Decision Regret Scale, will be compared between groups at baseline (T1) and in the week following the intervention (T2), one month and three months from baseline (T3 and T4). The decision regret scale is a five-item measure, on a scale from 1-5. Total scores will be added up, and higher scores represent greater decision regret. Lower scores represent less decision regret. The maximum score is 25 and the minimum score is 5.
Time Frame: At baseline (T1) and in the week following the intervention (T2), one month and three months from baseline (T3 and T4).
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Randomized Controlled Trial EMPOWER + Open Trial COVID-19 Phase Arm Combined | Randomized Controlled Trial Enhanced Usual Care Arm
Number analyzed (Participants) | 43 | 17
score on a scale
  Pre-Intervention Time 1 | 17.2 [10.3 to 24.1] | 19.4 [8.0 to 30.8]
  Post-Intervention Time 2 | 20.5 [15.3 to 25.6] | 15.3 [5.7 to 24.9]
  One Month Time 3 | 24.3 [19.1 to 29.5] | 18.5 [8.7 to 28.4]
  Three Months Time 4 | 19.1 [14.2 to 23.9] | 22.6 [13.7 to 31.6]

ADVERSE EVENTS:
Time Frame: 3 months
Description: For the purpose of this study, a Serious Adverse Event (SAE) is defined as an event that, as a direct result of the study, causes serious harm to the subject (e.g., that involvement in the study caused the death or serious injury to the subject).
Arm/Group | Randomized Controlled Trial EMPOWER Arm | Randomized Controlled Trial Enhanced Usual Care Arm | Open Trial COVID-19 Phase Arm
All-Cause Mortality (participants affected / at risk) | 0/18 | 0/17 | 0/25
Serious Adverse Events (participants affected / at risk) | 0/18 | 0/17 | 0/25
Other Adverse Events (participants affected / at risk) | 0/18 | 0/17 | 0/25

LIMITATIONS AND CAVEATS:
A caveat to the statistical analyses performed for this trial is that the original proposal assumed that there would be an "interventionist bias" for which we would need to adjust using approaches such as Hierarchical Linear Modeling (HLM). This resulted in a deviation from the original proposed use of HLM because there was no need to correct for clustering within interventionists.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-12-14): https://cdn.clinicaltrials.gov/large-docs/59/NCT03276559/Prot_SAP_001.pdf
  • Informed Consent Form (2023-09-18): https://cdn.clinicaltrials.gov/large-docs/59/NCT03276559/ICF_000.pdf